CLINICAL TRIAL: NCT01582035
Title: A Phase I, Open Label Trial in Genotype 1 HCV-Infected Subjects to Determine the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Repeated Doses of TMC647055 Given in Combination With Telaprevir
Brief Title: Study to Examine Multiple Doses of TMC647055 in Combination With Telaprevir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100735; TMC647055HPC1005 (Other: Janssen R&D Ireland); 2011-004028-37 (EudraCT Number)
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC647055HPC1005; TMC647055; telaprevir
MeSH Terms: conditions — Hepatitis C | interventions — 27-cyclohexyl-12,13,16,17-tetrahydro-22-methoxy-11,17-dimethyl-10,10-dioxide-2,19-methano-3,7:4,1-dimetheno-1H,11H-14,10,2,9,11,17-benzoxathiatetraazacyclo docosine-8,18(9H,15H)-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panel 1 (Experimental): TMC647055 in combination with TVR for 10 days. Immediately followed by the extension phase: TVR at a dose of 750 mg every 8 hours for 12 weeks in combination with Peg IFN and RBV followed by either 12 or 36 weeks of PegIFN -RBV treatment alone.
  Interventions: Drug: TMC647055; Drug: TVR; Drug: PegFN; Drug: RBV
- Panel 2 (Experimental): TMC647055 in combination with TVR for 10 or 14 days. Immediately followed by the extension phase: TVR at a dose of 750 mg every 8 hours for 12 weeks in combination with Peg IFN and RBV followed by either 12 or 36 weeks of PegIFN -RBV treatment alone.
  Interventions: Drug: TMC647055; Drug: TVR; Drug: PegFN; Drug: RBV

INTERVENTIONS:
Drug: TMC647055 — type=exact number, unit=mg, number=500, form=solution, route=oral use. Panel 1: TMC647055 is to be taken twice daily at a dose of 500 mg per day for 10 days.
  Arms: Panel 1
Drug: TMC647055 — type=exact number, unit= mg, number=up to macimum 1000, form=solution, route=oral use. Panel 2: TMC647055 is to be taken twice daily at a maximum dose of 1000 mg for 10 or 14 days.
  Arms: Panel 2
Drug: TVR — type=exact number, unit= mg, number=1125, form=tablet, route=oral use. TVR is to be taken twice daily at a dose of 1125 mg for 10 days.
  Arms: Panel 1
Drug: TVR — type=exact number, unit=mg, number=1125 or 1500, form=tablet, route=oral use. In panel 2: TVR is to be taken twice daily at a dose of 1125 or 1500 mg for 10 or 14 days. In panel 3: TVR is to be taken twice daily at a dose of 1125 or 1500 mg for 6 days with on day 6 a morning dose only.
  Arms: Panel 2
Drug: TVR — type= exact number, unit= mg, number=750, form=tablet, route=oral use. TVR is to be taken every 8 hours at a dose of 750 mg for 12 weeks.
Drug: PegFN — type= exact number, unit= mcg, number=180, form=solution, route=subcutaneous. PegIFN is to be injected once per week for 24 or 48 weeks.
Drug: RBV — type=exact number, unit=mg, number=1000 or 1200, form=tablet, route=oral use. RBV is to be taken at 1000 or 1200 mg per day in 2 divided doses, depending on the weight for 24 or 48 weeks.

SUMMARY:
The purpose of this study is to assess safety, tolerability, pharmacokinetics (how the drug is absorbed into the bloodstream) and antiviral activity of repeated doses of TMC647055 given in combination with telaprevir in HCV infected patients. TMC647055 is being investigated for the treatment of hepatitis C infection. Telaprevir has recently been approved in the USA and in Europe for the treatment of chronic hepatitis C infected patients.

DETAILED DESCRIPTION:
This is a phase I, open label trial in genotype 1 hepatitis C virus (HCV) infected patients. The study population consists of 16 adult patients. TMC647055 is given as an oral solution and telaprevir (TVR) is given as oral tablets. Patients found to be eligible after the screening visit will be divided over 2 panels that will be performed sequentially. In the first panel, 8 patients will receive TMC647055 at a dose of 500 mg twice a day in combination with TVR at a dose of 1125 mg twice a day for 10 consecutive days. In the second panel, 8 subjects will receive TMC647055 in combination with TVR for 14 days. TMC647055 and TVR dose will be decided based on results from panel 1. TMC647055 dose will not be higher than 1000 mg twice a day and TVR dose will be 1125 mg twice a day or 1500 mg twice a day. It could also be decided to change duration of panel 2 to 10 days. In that case, the timing of assessments of panel 1 will be followed. For the duration of dosing in the 2 panels, patients will remain on site. Immediately after the last dose in panels 1 and 2, patients will start the extension phase. In this phase, patients will receive TVR at a dose of 750 mg every 8 hours for 12 weeks in combination with pegylated interferon alfa (Peg IFN)(180ug subcutaneous once weekly) and ribavirin (RBV) (1000 or 1200 mg per day orally depending on weight in 2 divided doses). After that they will receive either 12 or 36 weeks of PegIFN -RBV treatment at the same dose regimen, depending on virus levels at week 4 and 12 in this extension phase. In the extension phase, patients will come to the site for visits at week 2, 4, 8, 12, 16, 24, 36 (if applicable) and 48 (if applicable). Patients who prematurely drop out in panel 1 or 2, will have a follow-up visit at 2 and 4 weeks after their last dose. Patients participating in the extension phase will have a follow-up visit at 4 and 12 weeks after their last dose. Safety and tolerability will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* genotype 1a or 1b HCV infection with HCV RNA level > 100,000 IU/mL
* A documented prior relapser patient to previous treatment regimens or treatment-naïve
* Patient must have documentation of a liver biopsy within 3 years before the screening visit or must agree to have a fibroscan/elastography examination within the screening period
* Patient is judged to be medically stable on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening

Exclusion Criteria:

* Evidence of liver cirrhosis
* Evidence of decompensated liver disease
* Evidence of any other cause of significant liver disease in addition to hepatitis C
* receiving or having received any treatment for HCV during the 6 months before screening
* History or evidence of current abuse of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise subject's safety and/or compliance with the study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Plasma PK parameters for TMC647055 and TVR after combination therapy in panel 1 and 2. | 9 samples at specific timepoints on days 1, 6 and 10 in panel 1, on days 1, 6 and 14 in panel 2 and daily on all other days in the 2 panels.
Number of participants with adverse events as a measure of safety and tolerability. | Continuously from screening until the last trial related visit.
Change from baseline values for clinical laboratory tests. | at screening, panel 1 on day 1, 6, 10 and 11, panel 2 on day 1, 6, 14 and 15, the 2 follow-up visits in case of drop-out from the panels, extension phase at every visit except the last follow-up visit
Change from baseline values for ECG and vital signs. | At screening, daily in panel 1 and 2 (Vital signs only in panel 1 day 1, 6, 11, in panel 2 day 1, 6, 15), at follow-up visits in case of drop-our from the panels, in extension phase at week 4, 12, 16 (ECG only), 24, 36, 48 and first follow-up visit
Change from baseline for physical examination. | at screening, panel 1 on day 1, 6 and 11, panel 2 on day 1, 6 and 15, extension phase at the week 4, 12, 24, 36, 48 and first follow-up visit
Individual evalution of HCV RNA levels. | For the 2 panels: 3 samples on day 1, 2 samples on day 2 and further daily samples except day 7 & 9 in panel 1 and day 7, 9, 11 & 13 in panel 2.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (2):
- Germany (2):
  - Berlin
  - München

REFERENCES:
- See also: A Phase 1, open-label trial in genotype 1 HCV infected subjects to determine the safety, tolerability, pharmacokinetics, and antiviral activity of repeated doses of TMC647055 given in combination with telaprevir — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3400&filename=CR100735_CSR.pdf